CLINICAL TRIAL: NCT00660244
Title: Breast Cancer Tumor Care Patient Observation Programme
Brief Title: Breast Cancer Tumor Care Observational Programme
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OAT-ARI-2007/1
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Post Menopausal; Arthralgia
Keywords: Arimidex; Post menopausal; arthralgia
MeSH Terms: conditions — Arthralgia | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole — Oral
  Other Names: Arimidex

SUMMARY:
The purpose of this study is to investigate efficacy and tolerability under anastrozole (Arimidex) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Already on upfront Arimidex Therapy (Start 1-4 weeks before)
* HR+

Exclusion Criteria:

* Premenopausal women
* Tamoxifen switch patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-02; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression of disease and tolerability in general | Baseline, every 3 month

SECONDARY OUTCOMES:
Patient questionnaire to collect data on Incidence, time of onset and treatment of arthralgia | Baseline, every 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Melichart, Study Chair — Hospital Rudolfstiftung; Dr. Feistauer, Study Chair — AKH-Vienna
Locations (1):
- Research Site, Graz, Austria